CLINICAL TRIAL: NCT03325543
Title: Can Women Correctly Contract Their Pelvic Floor Muscles After to Receive Verbal Instructions and Vaginal Palpation? Protocol of a Randomized Controlled Clinical Trial
Brief Title: Can Women Correctly Contract Their Pelvic Floor Muscles After to Receive Verbal Instructions and Vaginal Palpation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Letícia de Azevedo Ferreira, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2017-10-16; First posted 2017-10-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Urinary Incontinence; Urinary Incontinence, Stress; Urination Disorders; Lower Urinary Tract Symptoms
Keywords: Urinary Incontinence, Stress; Pelvic Floor; Exercise
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress; Urination Disorders; Lower Urinary Tract Symptoms; Motor Activity | interventions — Observation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: verbal instruction + body awareness techniques + vaginal palpation (Experimental): The intervention group will receive verbal instructions on the anatomy and function of PFMs associated with the use of body awareness techniques and vaginal palpation to learn the correct PFMs contraction. The intervention program will last four weeks, and will contain four outpatient consultations (1 session per week) lasting 60 minutes each session.
  Interventions: Other: Visual observation; Other: Vaginal palpation (bidigital touch)
- Control group: verbal instruction + body awareness techniques (Active Comparator): The control group will receive visual and verbal orientations of the anatomy and function of PFMs associated with the use of body awareness techniques and visual observation of the PFM.
  Interventions: Other: Visual observation

INTERVENTIONS:
Other: Visual observation — Verbal instructions about the anatomy, function and how to perform the pelvic floor muscle contraction
Other: Vaginal palpation (bidigital touch) — The physiotherapist touched the patients' perineal region (vulva, tendinous centre of the perineum and external region of the anal canal) with a spatula and asked them to identify the pointed region; and with the digital palpation, the physiotherapist touched the tendinous centre of the perineum, pressing it in the cranial direction, and instructed the patients to contract the pelvic floor muscle
  Arms: Experimental group: verbal instruction + body awareness techniques + vaginal palpation

SUMMARY:
The pelvic floor muscle training (PFMT) is a conservative treatment, currently considered as first line for women with stress urinary incontinence (SUI). However, in practice, about 30 to 50% of women are unable to perform the correct contraction of the pelvic floor muscles (PFMs). When requested to perform the muscle contraction, the contraction of the gluteal muscles, hip adductors, or abdominal muscles is observed initially, rather of contraction of the levator anus muscle. Some factors make it difficult to perform the contraction of the PFM, such as its location on the pelvic floor, and its small size, followed by a lack of knowledge of the pelvic region, as well as its functions. Associated with these factors is the use of the muscles adjacent to the PFM, as previously mentioned. In order for women to benefit from a PFMT program for the treatment of SUI, the awareness phase of PFM can't be omitted, since the literature is unanimous in stating that pelvic exercises improve the recruitment capacity of the musculature, its tone and reflex coordination during the effort activities.

DETAILED DESCRIPTION:
Research Questions: The objectives of this study is to test the hypothesis that the provision of verbal instructions about the anatomy and function of PFMs associated with the use of body techniques awareness and vaginal palpation helps in learning the correct contraction and improves the function of the PFMs.

Design: A single-centered, double-blind (investigator and outcome assessor) randomised controlled trial with two physiotherapy intervention groups.

Measurements: The primary outcome measure will be the number of fast muscle fibres, as determined by the number of effective contractions (fast and with full force contraction, 1 second each) out of ten contractions performed. The secondary outcome measure will be the PFM function (vaginal palpation and visual observation), the occurrence of associated contractions of the abdominal, gluteal and adductor muscles during the voluntary contraction of PFM , and self-efficacy scale for practising PFM exercises.

ELIGIBILITY:
Inclusion Criteria:

* Patients with predominance of SUI symptoms and ≥ 2 g leakage measured by pad test and without capability to contract the PFM properly

Exclusion Criteria:

* Not included if they were younger than 18 years old, had chronic degenerative diseases, pelvic organ prolapse greater than stage I by POP-Q, neurologic or psychiatric diseases, ability to contract PFMs, had previous pelvic floor re-education programs and/or pelvic floor surgeries

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2022-11-27 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Number of fast muscle fibres | After 4 weeks of supervised treatment
  Vaginal palpation (fast and with full force contraction, 1 second each)

SECONDARY OUTCOMES:
PFM function | After 4 weeks of supervised treatment
  Vaginal palpation
Occurrence of associated contractions | After 4 weeks of supervised treatment
  Contractions of the abdominal, gluteal and adductor muscles during the voluntary contraction of PFM
Self-perception of the effectiveness of perineal exercises will be evaluated by the Self-Efficacy Scale for Practice of Pelvic Floor Exercises | Questions about the expectation of results will be applied in the first week and after the fourth week of intervention.
  The scale is composed of 17 questions in the visual analogue scale format with responses ranging from 0 (not confident) to 100 (most confident). Thirteen questions refer to self-efficacy and four questions to expectation of results. The final result is obtained by averaging the items, which ranges from 0 to 100, where higher values are equivalent to more beneficial action of self-efficacy / expected result of the training of the PFM.

CONTACTS AND LOCATIONS:
Overall Officials: Letícia A Ferreira, Principal Investigator — Federal University of São Paulo
Locations (1):
- Letícia de Azevedo Ferreira, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Azevedo Ferreira L, Fitz FF, Gimenez MM, Matias MMP, Bortolini MAT, Castro RA. The role of vaginal palpation in motor learning of the pelvic floor muscles for women with stress urinary incontinence: study protocol for a randomized controlled trial. Trials. 2020 Jul 31;21(1):693. doi: 10.1186/s13063-020-04624-4. PMID 32736576